CLINICAL TRIAL: NCT02113527
Title: Evaluation of Gastric Emptying Time, Gastric Electrical Activity and Gastrointestinal Peptides to Identify Dyspeptic Patients With Epigastric Pain Syndrome From Those With Postprandial Distress Syndrome According to the Rome III Proposed Subdivision of Functional Dyspepsia
Brief Title: Gastric Activity and Gastrointestinal Peptides in Patients With Functional Dyspepsia
Acronym: DYSMOT-RIII
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Francesco Russo, Senior researcher, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: RC192014
Record Dates: First submitted 2014-03-26; First posted 2014-04-14 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Dyspepsia
Keywords: Electrogastrography; Functional dyspepsia; Gastric emptying; Gastrointestinal peptides; Rome III criteria
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — breath specimen, whole blood, serum, white cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Epigastric pain syndrome (EPS): Patients suffering from functional dyspepsia characterized by epigastric pain syndrome according to Rome III criteria
- Postprandial distress syndrome (PDS): Patients suffering from functional dyspepsia characterized by postprandial distress syndrome according to Rome III criteria
- Healthy subjects: Healthy subjects as control group

SUMMARY:
Rome III criteria defined functional dyspepsia (FD) as the presence of symptoms from the gastroduodenal region in the absence of any organic, systemic or metabolic disease that is likely to explain the symptoms. FD can be further subdivided into two diagnostic categories: postprandial distress syndrome (PDS) and epigastric pain syndrome (EPS).

Disorders of gastric electric activity and abnormal gastric emptying are probably actively involved in the FD onset. Different noninvasive procedures may be applied in order to evaluate the gastric motor functions such as 13C breath testing and cutaneous electrogastrography. Besides, different gastrointestinal peptides (i.e. CCK, peptide YY, Neurotensin, Somatostatin, Leptin, Ghrelin, Motilin, Gastrin, Pepsinogen I and II) are involved in the control of gastroduodenal motility.

Aims of the present study are: 1) to evaluate the GI peptide circulating concentrations, the gastric electrical activity and gastric emptying time by applying noninvasive procedures in patients suffering from functional dyspepsia and 2) to test whether a significant difference exists between the two diagnostic categories of meal-induced dyspeptic symptoms

DETAILED DESCRIPTION:
Functional dyspepsia is one of the most relevant functional gastrointestinal disorders (FGIDs) among general population. Rome III criteria defined functional dyspepsia as the presence of symptoms from the gastroduodenal region (early satiation, postprandial fullness, epigastric pain or burning) in the absence of any organic, systemic or metabolic disease that is likely to explain the symptoms. Etiological causes are still unclear, and the pathophysiological mechanisms still largely unknown. Besides, Helicobacter pylori infection is often present in these patients and contributes to complicate the clinical presentation. One of the main problem in the management of these patients is the lack of reliable biohumoral markers. Thus, functional disorders are usually diagnosed on the bases of symptomatic patterns. The Rome consensus has proposed to further subdivide FD into two diagnostic categories of meal-induced dyspeptic symptoms: postprandial distress syndrome (PDS), characterized by postprandial fullness and early satiation, and epigastric pain syndrome (EPS), characterized by epigastric pain and burning.

Central processing of visceral stimuli, and its role in the pathogenesis of functional dyspepsia, as well as low-grade inflammation in the duodenum are important emerging topics in pathophysiology research. In this framework, disorders of gastric electric activity and abnormal gastric emptying are probably actively involved in the onset of symptomatology. Different noninvasive procedures may be applied in order to evaluate the gastric motor functions. Among them, gastric emptying time evaluation by 13C breath testing and cutaneous electrogastrography have raised attention for their reliability and potentiality. Another important pathophysiological concern of FD is represented by the possible alterations in circulating concentrations of different gastrointestinal peptides at various degree involved in the control of gastroduodenal motility [namely Cholecystokinin (CCK), peptide YY, Neurotensin, Somatostatin, Leptin, Ghrelin, Motilin, Gastrin, Pepsinogen I and II]. In previous studies significant lower levels of motilin was found in dyspeptic patients with altered antroduodenal motility was found. CCK mediates satiety by acting on the CCK receptors distributed widely throughout the central nervous system as well as effects on the vagus nerve. Other experimental data suggest that somatostatin and neurotensin may affect muscle contractility and delay the intestinal transit.

On these bases aims of the study will be: 1) to evaluate the GI peptide circulating concentrations, the gastric electrical activity and gastric emptying time by applying noninvasive procedures in patients suffering from functional dyspepsia and 2) to test whether a significant difference exists between the two diagnostic categories of meal-induced dyspeptic symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from dyspeptic symptoms according to Rome III;
* Helicobacter pylori negative subjects;
* age 19-70 yr.;
* willingness to complete the study;
* not recent administration (in the 2 months before the examination) of anti-inflammatory drugs (NSAIDs), antibiotics, bismuth, antacids, H2-receptor antagonists, proton pump inhibitor, sucralfate or misoprostol;
* at least one endoscopic/radiological GI evaluation in the last 5 yrs.

Exclusion Criteria:

* previous history of gastric tumors or gastric surgery
* lactose intolerance;
* celiac disease, wheat sensitivity;
* alarm symptoms (GI bleeding, weight loose etc.);
* psychiatric diseases;
* familial history of peptic ulcer;
* gastric cancer or IBD;
* abnormal thyroid function;
* other exclusion criteria (namely, pregnancy, breast-feeding, and drug allergies).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in this observational study from the out-patients of the National Institute of Digestive Diseases, I.R.C.C.S. Saverio de Bellis, Castellana Grotte, Bari, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Fasting plasma concentration of GI peptides, gastric emptying time and dyspepsia subtype. | Duration of 4-hour study visit
  Exploration of relationships between GI peptide concentrations (CCK, peptide YY, Neurotensin, Somatostatin, Leptin, Ghrelin, Motilin, Gastrin, Pepsinogen I and II), solid gastric emptying, and dyspepsia subtype.
  Blood samples will be compared pre/post test meal for FD cohorts (EPS/PDS) and controls: 0 time/baseline and 16 times/post meal.
  Associations of plasma GI peptides pre and postprandial levels & gastric emptying will be studied.
  Amount of 13CO2 will be determined for each time point (1 pre/ 16 post meal) using equation nested in software package with IRMS.
  The concentration of 13CO2 and 12CO2 in the exhaled breath samples will be measured by mass spectrometry.

SECONDARY OUTCOMES:
Gastric electrical activity and GI peptides according functional dyspepsia subtype | Duration of 4-hour study visit
  Correlations between plasma GI peptide concentrations and gastric electrical activity to be measured during gastric emptying time evaluation.
  Gastric electrical activity will be measured by cutaneous electrogastrography.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Russo, MD, Principal Investigator — IRCCS "S. de Bellis"
Locations (1):
- National Institute of Digestive Diseases IRCCS "Saverio de Bellis", Castellana Grotte, Bari, Italy

REFERENCES:
- [Background] Chasen M, Bhargava R. Gastrointestinal symptoms, electrogastrography, inflammatory markers, and PG-SGA in patients with advanced cancer. Support Care Cancer. 2012 Jun;20(6):1283-90. doi: 10.1007/s00520-011-1215-8. Epub 2011 Jun 19. PMID 21688162
- [Background] Miwa H, Watari J, Fukui H, Oshima T, Tomita T. [Pathogenesis and management of functional dyspepsia]. Nihon Rinsho. 2010 Jul;68(7):1391-401. Japanese. PMID 20662226
- [Background] Khoo J, Rayner CK, Feinle-Bisset C, Jones KL, Horowitz M. Gastrointestinal hormonal dysfunction in gastroparesis and functional dyspepsia. Neurogastroenterol Motil. 2010 Dec;22(12):1270-8. doi: 10.1111/j.1365-2982.2010.01609.x. Epub 2010 Oct 5. PMID 20939851
- [Background] De Smet B, Mitselos A, Depoortere I. Motilin and ghrelin as prokinetic drug targets. Pharmacol Ther. 2009 Aug;123(2):207-23. doi: 10.1016/j.pharmthera.2009.04.004. Epub 2009 May 6. PMID 19427331
- [Background] Geeraerts B, Mimidis K, van Oudenhove L, Vos R, Karamanolis G, Tack J. Role of endogenous opioids in the control of gastric sensorimotor function. Neurogastroenterol Motil. 2008 Oct;20(10):1094-102. doi: 10.1111/j.1365-2982.2008.01144.x. Epub 2008 May 15. PMID 18482249